CLINICAL TRIAL: NCT06386744
Title: Pilot Study of SGX945 (Dusquetide) in the Treatment of Aphthous Ulcers in Behcet's Disease
Brief Title: Dusquetide for the Treatment of Behcet's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Soligenix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DUS-AUBD-01
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Behçet Disease
Keywords: dusquetide
MeSH Terms: conditions — Behcet Syndrome | interventions — dusquetide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SGX945 (Experimental): This is an open-label study and all participants will receive SGX945.
  Interventions: Drug: Dusquetide

INTERVENTIONS:
Drug: Dusquetide — 1.5 mg/mL dusquetide administered as a 4 minute IV infusion, twice per week for 4 weeks
  Other Names: SGX945; SGX942

SUMMARY:
This is a clinical study to see if dusquetide can treat flares of oral and genital ulcers caused by Behcet's Disease. Study participants will receive an infusion of dusquetide twice a week for 4 weeks (8 treatments total), with weekly follow-up visits for an additional 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a clinical diagnosis of Behcet's Disease meeting the International Study Group criteria.
* Participants must have at least two oral ulcers and/or one genital ulcer on the day of randomization.
* Participants willing to follow the clinical protocol and voluntarily give their written informed consent.
* Female participants not pregnant or nursing and willing to undergo a pregnancy test prior to treatment initiation and at the end of the treatment period.

Exclusion Criteria:

* Pregnancy or mothers who are breast-feeding.
* All women of childbearing potential (WOCBP) and males with female partners who are WOCBP not willing to agree to the use of effective contraception during the trial.
* Evidence of significant renal, hepatic, hematologic or immunologic disease.
* Use of any investigational medication within 4 weeks prior to enrollment or 5 pharmacokinetic/pharmacodynamic half-lives (whichever is longer).
* Having received concomitant immune modulating therapy (except colchicine or azathioprine) within:

  1. Ten days prior to enrollment for mycophenolate mofetil
  2. Four weeks (28 days) prior to enrollment for cyclosporine, methotrexate, cyclophosphamide, thalidomide and dapsone
  3. Oral and topical corticosteroids must have been tapered as appropriate and discontinued 3 days prior to day of enrollment
  4. At least 5 terminal half-lives for all biologics including, but not limited to, those listed below; within: i. Four weeks prior to enrollment for etanercept; ii. Eight weeks prior to enrollment for infliximab; iii. Ten weeks prior to enrollment for adalimumab, golimumab, certolizumab, abatacept, and tocilizumab; iv. Six months prior to enrollment for secukinumab.
* Having received oral or parenteral corticosteroids within 6 weeks (42 days) prior to enrollment.
* Having received apremilast (Otezla) within 4 weeks prior to enrollment.
* Presence of non- Behcet's Disease related genital ulcers, including both infectious and non-infectious etiologies.
* Active organ involvement requiring immunosuppressive treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Number of Oral Ulcers | 4 weeks
  The number of oral ulcers will be counted at baseline and each visit during the treatment period.
Number of Genital Ulcers | 4 weeks
  The number of genital ulcers will be counted at baseline and each visit during the treatment period.

SECONDARY OUTCOMES:
Pain of Oral Ulcers | 4 weeks
  The pain of oral ulcers will be measured using a 10 cm Visual Analog Scale (VAS) at baseline and each visit during the treatment period.
Pain of Genital Ulcers | 4 weeks
  The pain of genital ulcers will be measured using a 10 cm Visual Analog Scale (VAS) at baseline and each visit during the treatment period.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University - Cerrahpasa, Cerrahpasa School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Donini O, Sulu B, Pullion C, Rumage A, Straube R, Schaber C, Hatemi G. Results from a pilot study of dusquetide for the treatment of aphthous ulcers associated with Behcet syndrome. Rheumatology (Oxford). 2025 Dec 16:keaf682. doi: 10.1093/rheumatology/keaf682. Online ahead of print. PMID 41400947